CLINICAL TRIAL: NCT04238650
Title: A Randomised, Double Blind, Two-Arm, Single Dose, Parallel Phase I Study To Compare the Pharmacokinetics, Safety and Immunogenicity of MB02 (a Proposed Bevacizumab Biosimilar Drug) and EU Approved Avastin® in Japanese Healthy Male Volunteers
Brief Title: A Pharmacokinetic Study Comparing MB02 And EU Avastin® In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: mAbxience Research S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MB02 A 04-18
Record Dates: First submitted 2020-01-16; First posted 2020-01-23 (Actual); Results first posted 2021-02-01 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Healthy Volunteers; Male; Japanese

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB02 (Bevacizumab Biosimilar) (Experimental): Intervention Description: Sterile vial 400mg/16ml, single-dose 3mg/kg administered as 90-minute infusion on day 1.
  Interventions: Drug: MB02 (Bevacizumab Biosimilar)
- EU approved Avastin® (Active Comparator): Intervention Description: Sterile vial 400mg/16ml, single-dose 3mg/kg administered as 90-minute infusion on day 1.
  Interventions: Drug: EU approved Avastin®

INTERVENTIONS:
Drug: MB02 (Bevacizumab Biosimilar) — Solution for intravenous infusion, single dose of 3mg/kg, administered as 90- minute infusion
  Arms: MB02 (Bevacizumab Biosimilar)
Drug: EU approved Avastin® — Solution for intravenous infusion, single dose of 3mg/kg, administered as 90- minute infusion
  Arms: EU approved Avastin®

SUMMARY:
A Randomised, Double Blind, Two-Arm, Single Dose, Parallel Phase I Study To Compare the Pharmacokinetics, Safety and Immunogenicity of MB02 (a Proposed Bevacizumab Biosimilar Drug) and EU Approved Avastin® in Japanese Healthy Male Volunteers.

During the course of the study, the similarity in pharmacokinetics will be assessed by sampling the levels of drug in the blood, and by comparing these levels among the different administration arms. Safety, tolerability, and immunologic response to the administered drugs will also be evaluated throughout.

DETAILED DESCRIPTION:
The primary PK parameter endpoint is AUC(0-∞) for bevacizumab. The secondary PK endpoints will include all other PK parameters for bevacizumab, including Cmax, tmax, t1/2, CL and AUClast.

The serum PK parameters of bevacizumab will be calculated using standard noncompartmental methods. An analysis of covariance model will be used to analyse the log-transformed primary PK parameters (AUC[0-∞] and Cmax) and AUClast. The model will include a fixed effect for treatment and body weight as a covariate.

All other PK parameters will not be subject to inferential statistical analysis.

Estimates of geometric mean ratios together with the corresponding 90% confidence intervals (CI) will be derived for the comparisons of the PK parameters as follows:

• MB02 versus EU Avastin®

A mixed effects model with treatment arm as fixed effect will be used to compare natural-logarithmic transformed PK parameters (AUC[0-∞+, AUClast and Cmax) between the two treatment arms (MB02 vs EU-approved Avastin®)

PK similarity between arms will be concluded if the 90% confidence intervals (CIs) for the geometric mean test/reference ratio of AUC(0-∞) fell within the predefined 0.80-1.25 bioequivalence interval.

All AEs will be listed and summarised using descriptive methodology. All observed or patient-reported AEs will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The incidence of AEs for each treatment will be presented by severity and by association with the study drugs as determined by the Investigator (or designee). Each AE will be coded using the Medical Dictionary for Regulatory Activities. All safety data will be listed and summarised as appropriate.

Immunogenicity data (overall ADA incidence and titers, and neutralising ADA results) will be listed. A summary of the number and percent of subjects testing positive for ADA or neutralising antibodies before the dose of MB02, EU Avastin® (Day -1) and at scheduled post-dose assessments will be presented by treatment arm. All safety data and immunogenicity data summaries will be based on the safety analysis population. Select analyses may be repeated for subsets with or without ADA and de novo ADA formation as appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions. Subjects must have signed an informed consent before any study-related procedure or evaluation is performed.
2. Healthy Japanese males aged ≥20 to ≤55 years, inclusive, at Screening.
3. Subjects with Body mass index (BMI) between ≥18.5 to ≤28 kg/m2 and total body weight between ≥50 and ≤100 kg, at Screening
4. Subject must have no clinically relevant abnormalities identified by a detailed medical history.
5. Systolic blood pressure ≤140 mm Hg and diastolic blood pressure ≤90 mm Hg.
6. Computerized (12-lead) electrocardiogram (ECG) recording without signs of clinically relevant pathology.
7. All other values for hematology, coagulation and for biochemistry and urinalysis tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the Investigator, according to the following laboratory values:

   Adequate bone marrow function
   * Absolute neutrophil count ≥1.5 × 109 L
   * Platelet count ≥100 × 109 L
   * Hemoglobin >10 g/dl

   Adequate liver function:
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ ULN
   * Alkaline phosphatase (ALP) ≤1.5 × ULN
   * Total bilirubin <1.5 × ULN
   * Serum albumin: >3.5 g/dL
   * Low density lipoprotein cholesterol ≤139 mg/dL
   * High density lipoprotein cholesterol ≥ 40 mg/dL
   * Creatine kinase (CK) <2 ULN at D-1

   Adequate coagulation:

   • International normalised ratio (INR) 0.8 to 1.3

   Adequate renal function:
   * Blood urea nitrogen: ≤1.5 × ULN
   * Creatinine: <1.5 mg/dL
   * Urine dipstick for proteinuria <2+.
8. All intermittent medications should have been stopped at least 30 days prior to admission to the clinical research center.
9. Subjects agree to use contraception.
10. Ability and willingness to abstain from alcoholic beverages (alcohol) 48 hours prior to admission to the clinical research center.

Exclusion Criteria:

1. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients).
2. Previous treatment with an anti VEGF antibody like bevacizumab or any other protein or antibody targeting the VEGF receptor.
3. History of bleeding disorders or protein C, protein S, and/or factor V Leiden deficiency.
4. Known history of clinically significant essential hypertension (subjects under any antihypertensive treatment included), orthostatic hypotension, fainting spells or blackouts for any reason, cardiac failure or history of thromboembolic conditions.
5. History of GI perforation, ulcers, gastro oesophageal reflux, inflammatory bowel disease, diverticular disease, diverticular disease, any fistulae, pulmonary hemorrhage (hemoptysis) or reversible posterior leukoencephalopathy syndrome.
6. Any out-of-range laboratory values considered clinically significant by the investigator.
7. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
8. Any current or recent history of active infections, including localized infections. (Within 2 months prior Screening Visit for any serious infection which requires hospitalization or intravenous anti-infective, and within 14 days prior Screening Visit for any active infection which requires oral treatment). A negative result for human immunodeficiency virus (HIV), Hepatitis B (Hep B), and hepatitis C (Hep C) is required for participation. If subject shows positive Hepatitis B test, but results are compatible with prior immunisation and not infection may be included at the discretion of the Investigator.
9. Clinically relevant history of alcoholism, addiction or drug/chemical abuse prior to Check-in, and/or positive urinary drug test screen and/or positive breath alcohol test at Screening or Check in. Average intake of more than 24 units of alcohol / wk. (1 unit of alcohol equals ~250mL of beer, 100mL of wine or 35mL of spirits). Positive urine drug screen (opiates, methadone, cocaine, amphetamines (including ecstasy or methamphetamines), cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants and phencyclidine).
10. Treatment with non-topical medications within 7 days prior to study drug administration, with the exception of hormonal contraceptives, multivitamins, vitamin C, food supplements and a limited amount of acetaminophen, which may be used throughout the study.
11. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 60 days prior to Check-in, or within 5 half lives of the investigational drug used in the study.
12. Subjects considered unsuitable for inclusion by the investigator (e.g., inability to understand and comply with the study requirements or presence of any condition which, in the opinion of the investigator, would not allow safe participation in the study).
13. Strenuous exercise within seven days prior to admission to the clinical research center.
14. Significant or acute illness within 15 days prior to drug administration that may impact safety assessments per the judgement of the investigator.
15. Unsuitable veins for infusion and/or venepuncture.
16. History of, or planned surgery, including suturing, dental surgery or wound dehiscence within 30 days of dosing, or within 30 days of the last study visit. Presence of a nonhealing wound or fracture.
17. Medically significant dental disease or dental neglect with signs and or symptoms of local or systemic infection that would likely require a dental procedure during the course of the study.
18. Use or intend to use slow-release medications/products considered to still be active within 30 days prior to Check-in, unless deemed acceptable by the Investigator (or designee).
19. Have received a live or attenuated vaccine from 3 months prior to Screening or have the intention to receive a vaccine during the study.
20. Intend to travel to a region where a vaccination will be required due to endemic disease within 3 months of dosing.
21. Use of tobacco- or nicotine-containing products within 1 year prior to Check-in, or positive cotinine test upon Screening or Check-in.
22. Receipt of blood products within 60 days prior to Check-in.
23. Person who performed blood sampling more than 400 mL within 90 days before administration of investigational drug, more than 200 mL blood within 30 days, or blood donation of blood plasma / platelet component within 14 days.
24. History of abnormal peripheral sensation including paraesthesia and/or numbness in arms and/or legs.
25. Have previously received Bevacizumab either under present study or under any other circumstances.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only Japanese male subjects may be enrolled
Enrollment: 49 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2019-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi ETO, MD, Principal Investigator — SOUSEIKAI Hakata Clinic
Locations (1):
- SOUSEIKAI Hakata Clinic, Fukuoka, Japan

REFERENCES:
- [Derived] Eto T, Karasuyama Y, Gonzalez V, Del Campo Garcia A. A randomized, single-dose, pharmacokinetic equivalence study comparing MB02 (proposed biosimilar) and reference bevacizumab in healthy Japanese male volunteers. Cancer Chemother Pharmacol. 2021 Oct;88(4):713-722. doi: 10.1007/s00280-021-04324-z. Epub 2021 Jul 16. PMID 34269848

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 49 subjects were randomized and assigned to one of the study groups (24 to the MB02 arm and 25 to the EU Avastin arm). One subject that was randomized to EU Avastin® withdrew before receiving any study drug dose. Therefore, 48 subjects started the study treatment.
Period: Overall Study
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin®
Started | 24 | 25 (One subject was enrolled and randomized to EU Avastin® but the subject was not dosed (subject withdrawal before study drug administration))
Completed | 24 | 24
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin® | Total
Number analyzed (Participants) | 24 | 24 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (5.9) | 28.5 (6.6) | 28.4 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 24 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 24 | 24 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 67.0 (9.48) | 68.5 (9.13) | 67.75 (9.24)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.54 (2.26) | 23.33 (2.84) | 22.94 (2.57)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to Infinity [AUC(0-∞)]
Description: To compare the pharmacokinetic (PK) profiles of MB02 and EU Avastin® (in terms of AUC(0-∞)]) in Japanese population to establish bioequivalence between the 2 study drugs.
Time Frame: Predose, end of infusion, 2, 3, 4, 5, 6, 8, 12, 24 h post-dose on Day 1-8, Day 10, Day 14, Day 21, Day 28, Day 38, Day 50, Day 62, and Day 70.
Population: Overall number of participants analyzed equals to number of subjects who contributed to summary statistics.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin®
Number analyzed (Participants) | 24 | 24
ng*h/mL | 30200000 (14.7) | 29000000 (10.8)
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar) vs EU Approved Avastin®; Test type: Equivalence — Two treatments are judged not to be different from one another if the 90% CI of the ratio of a log-transformed exposure measure (AUC) falls completely within the range 0.80-1.25. The PK parameter AUC[0-∞] was log-transformed (base e) prior to analysis and was analysed using an ANCOVA model. The model included treatment as a fixed effect and body weight as a covariate; Ratio of GLSM = 1.04, 90% CI 2-sided [0.981 to 1.11]

2. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: To evaluate and compare the Cmax of MB02 and EU Avastin® in Japanese population.
Time Frame: as for outcome 1
Population: Overall number of participants analyzed equals to number of subjects who contributed to summary statistics.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin®
Number analyzed (Participants) | 24 | 24
ng/mL | 92900 (22.1) | 82300 (16.9)
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar) vs EU Approved Avastin®; Test type: Equivalence — Two treatments are judged not to be different from one another if the 90% CI of the ratio of a log-transformed exposure measure (Cmax) falls completely within the range 0.80-1.25. The PK parameter Cmax was log-transformed (base e) prior to analysis and was analysed using an ANCOVA model. The model included treatment as a fixed effect and body weight as a covariate; Ratio of GLSM = 1.13, 90% CI 2-sided [1.03 to 1.24]

3. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Observable Concentration (AUClast)
Description: To evaluate and compare the AUClast of MB02 and EU Avastin® in Japanese population.
Time Frame: as for outcome 1
Population: Overall number of participants analyzed equals to number of subjects who contributed to summary statistics.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin®
Number analyzed (Participants) | 24 | 24
ng*h/mL | 28200000 (12.3) | 26800000 (9.18)
Statistical Analysis 1: Comparison: MB02 (Bevacizumab Biosimilar) vs EU Approved Avastin®; Test type: Equivalence — Two treatments are judged not to be different from one another if the 90% CI of the ratio of a log-transformed exposure measure (AUC) falls completely within the range 0.80-1.25. The PK parameter AUClast was log-transformed (base e) prior to analysis and was analysed using an ANCOVA model. The model included treatment as a fixed effect and body weight as a covariate; Ratio of GLSM = 1.05, 90% CI 2-sided [0.997 to 1.11]

4. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax)
Description: To evaluate and compare the tmax of MB02 and EU Avastin® in Japanese population.
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin®
Number analyzed (Participants) | 24 | 24
h | 4.50 [1.52 to 24.00] | 4.00 [1.52 to 12.00]

5. Secondary Outcome: Apparent Serum Terminal Elimination Half Life (t1/2)
Description: To evaluate and compare the t1/2 of MB02 and EU Avastin® in Japanese population.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin®
Number analyzed (Participants) | 24 | 24
h | 430 (16.4) | 450 (12.9)

6. Secondary Outcome: Total Body Clearance (CL)
Description: To evaluate and compare the CL of MB02 and EU Avastin® in Japanese population.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin®
Number analyzed (Participants) | 24 | 24
L/h | 0.00660 (18.3) | 0.00702 (14.4)

7. Secondary Outcome: Volume of Distribution (Vz)
Description: To evaluate and compare the Vz of MB02 and EU Avastin® in Japanese population.
Time Frame: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin®
Number analyzed (Participants) | 24 | 24
L | 4.10 (13.2) | 4.56 (12.5)

8. Secondary Outcome: Incidence of Treatment-related Adverse Events (Safety)
Description: Compare the incidence of TEAEs reported in each treatment arm using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Time Frame: Day 1 - Day 70
Population: TEAEs were assessed in the Safety population. Subjects receiving MB02 or EU Avastin® and with at least 1 post-dose safety assessment comprised the Safety population.
Measure: Number; unit: participants
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin®
Number analyzed (Participants) | 24 | 24
participants
  Subjects with TEAEs | 8 | 12
  TEAEs of mild severity | 8 | 9
  TEAEs of moderate severity | 2 | 6
  TEAEs of severe severity | 0 | 0
  Related TEAEs | 0 | 2
  Subjects with SAEs | 0 | 0
  Subjects discontinued due to TEAEs | 0 | 0

9. Secondary Outcome: Incidence of ADA Including Nab (Immunogenicity)
Description: Incidence of anti-bevacizumab antibodies (ADA), including neutralizing antibodies (Nab). Subjects who tested positive at baseline are not included here.
Time Frame: Day -1, Day 14, 28, 50 and 70.
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin®
Number analyzed (Participants) | 24 | 24
participants
  ADA positive | 0 | 1
  nAb positive | 0 | 1
  NO seroconversion | 24 | 23

ADVERSE EVENTS:
Time Frame: Day 1-Day 70
Description: Coded according to Medical Dictionary for Regulatory Activities (version 22.1), and graded on the basis of the US National Cancer Institute's Common Terminology for Adverse Events (version 5.0).
  For the purpose of safety reporting in healthy volunteers, all serious adverse events were considered unexpected and reported as suspected unexpected adverse reactions (SUSARs).
Arm/Group | MB02 (Bevacizumab Biosimilar) | EU Approved Avastin®
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 8/24 | 12/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MB02 (Bevacizumab Biosimilar) (N=24) | EU Approved Avastin® (N=24)
Nasopharyngitis (Infections and infestations) | 2 (2) | 6 (6)
Pharyngitis (Infections and infestations) | 1 (1) | 4 (5)
Blood Creatine Phosphokinase Increased (Investigations) | 3 (4) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 2 (3) | 2 (2)
Aspartate Aminotransferase Increased (Investigations) | 2 (3) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results.

DOCUMENTS (2):
  • Study Protocol (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT04238650/Prot_002.pdf
  • Statistical Analysis Plan (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/50/NCT04238650/SAP_003.pdf